CLINICAL TRIAL: NCT05626582
Title: Effects of Acute Pain vs Context Change on Motor Learning Retention in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Susanne M Morton, Associate Professor, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1786370-1.3; R01AG071585 (NIH)
Record Dates: First submitted 2022-11-13; First posted 2022-11-23 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Pain, Acute; Motor Activity
Keywords: acute pain; young adults; pain; motor learning; motor consolidation; gait; locomotion; walking; generalization
MeSH Terms: conditions — Acute Pain; Motor Activity; Pain

STUDY DESIGN:
Masking Description: Application of pain or no stimulus cannot be masked from participants, nor from outcomes assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pain Stimulus - Learning Only (Experimental): Capsaicin combined with heat applied to intact skin
  Interventions: Procedure: pain delivery - learning only
- Pain Stimulus - Learning and Retention (Experimental): Capsaicin combined with heat applied to intact skin
  Interventions: Procedure: pain delivery - learning and retention
- No Stimulus (No Intervention): Nothing applied to skin

INTERVENTIONS:
Procedure: pain delivery - learning only — Experimental pain paradigm delivered (capsaicin cream combined with heat) that is short-term and painful but not harmful. Applied to skin just during the Day 1 learning period.
  Arms: Pain Stimulus - Learning Only
Procedure: pain delivery - learning and retention — Experimental pain paradigm delivered (capsaicin cream combined with heat) that is short-term and painful but not harmful. Applied to skin during the Day 1 learning period and again during the Day 2 retention period.
  Arms: Pain Stimulus - Learning and Retention

SUMMARY:
To date, the effects of pain on motor learning have not been thoroughly investigated. When examining potential effects on retention of motor learning, it is important to dissociate any effects of pain from effects of a context change. The purpose of this research is to determine whether any altered retention of motor learning associated with acute pain is a true affect of pain or an affect of context (or both).

ELIGIBILITY:
Abbreviations: HR= heart rate, bpm= beats per minute; BP= blood pressure; ADD= attention deficit disorder; ADHD= attention deficit hyperactivity disorder; MoCA= Montreal Cognitive Assessment; GAD-7= Generalized Anxiety Disorder 7 Scale; PHQ-2, PHQ-9= Patient Health Questionnaire-2 and -9.

Inclusion Criteria:

* 18-35 years old
* Self-identifying as generally medically healthy
* Able to read, write and speak English
* Able to provide informed consent
* Willing to undergo the experimental pain or non-painful electrical stimulation, if selected

Exclusion Criteria:

* Resting HR < 50 or > 100 bpm
* Resting BP < 90/60 or > 140/95 mmHg
* Any history or current mental health condition, learning/developmental disability or cognitive impairment, including ADD/ADHD, severe anxiety, severe depression, autism spectrum disorder, insomnia, mild cognitive impairment, etc.
* Score on the MoCA <23
* Score on the GAD-7 ≥ 10
* Score on the PHQ-2 ≥ 2 and score on the PHQ-9 ≥ 10
* Any current (within last 3 month) or chronic medical conditions, including any musculoskeletal, cardiovascular, endocrine, pulmonary, metabolic, psychiatric or neurological diagnosis
* Any implanted electronic medical devices (i.e., cardiac pacemakers, cardiac defibrillators, spinal cord neurostimulators)
* Any impaired sensation or weakness in either lower extremity or in the area targeted for the stimulus
* History of serious concussion or head injury, defined as a loss of consciousness for > 5 minutes and/or requiring medical treatment, or > 2 concussions over the lifespan
* Any history of acute or chronic problems with balance, any dizziness, or > 1 fall in the last 12 months
* Taking 4 or more medications
* Currently or regularly using any analgesic medications, over-the-counter remedies, or any other treatment for the purposes of pain relief (i.e., baby aspirin for heart health permitted, etc.)
* Any current or chronic pain condition during the last year, located anywhere in the body
* Allergy to capsaicin or hot peppers
* Any skin lesion, breakage or irritation in the area targeted for the painful stimulus
* Skin sensitivity to soaps/creams/perfumes or to heat
* Poor circulation in the area targeted for the painful stimulus
* Prior participation in a locomotor learning study in this lab within the last 2 years

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Motor Retention Magnitude | 24 hours post learning (day 2)
  degree to which the learned locomotor pattern has been remembered (in step length percent change, normalized to the amount learned from day 1)
Motor Learning Magnitude | immediately after learning (day 1)
  degree to which the new locomotor pattern has been acquired (in step length percent change)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne M Morton, PhD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States